# INFORMED CONSENT FORM

Online Training to Improve Evidence-based Leadership
Competencies Among Nurse Leaders in China: Study
Protocol for a Randomised Feasibility Trial
(EVILEAD-CH)

NCT number: NCT05244499

Date of the document: 15 February 2023

#### INFORMED CONSENT FORM

- 1. Project Title: Leadership training to improve the evidence-based leadership competencies of nursing leaders
- 2. Principal investigators: Xianhong LI PhD, professor, Xiangya School of Nursing, Central South University; VÄLIMÄKI Maritta PhD, Professor, University of Turku

You are invited to participate in the research program titled Leadership training to improve the evidence-based leadership competencies of nursing leaders, which aims to provide references for intervention development for enhancing the evidence-based leadership of nursing leaders.

The project will be from August 2022 to February 2023, seven months in total.

If you agree to participate in the project:

- 1. You will be interviewed by the principal investigators at a date and time convenient to you.
- 2. You may be asked questions about the number of times you have participated in the project, your perceptions, etc., one week after the termination of the project in an audio-recorded interview that will last approximately 30 minutes.
- 3. You will be asked to fill in a questionnaire survey (three times in total, before the project, right after the project, and 7 months after the project)
- 4. You can withdraw from the study at any time for any reason.
- 5. After the interview, you will receive a bookmark as a gift for participation.

If you are in Group A, you will register on the Xiaoetong online learning platform after signing the informed consent and participate in a 7-month evidence-based leadership training program. The program will consist of 7 recorded online modules, and we will conduct one module per month. Each module will focus on one topic and last around 30 minutes. After the online modules, there will be post-module tasks and/or reading materials (e.g., PowerPoint, literature, videos). Participants are required to finish the post-module tasks and upload them to the online platform before the next module. Participants can choose their study time within the time period specified by researchers. For example, the task for the first module is to identify a leadership issue that the participants face in their daily work, describe it clearly, and then upload the detailed (leadership) issue to the learning platform before the next module initiates. The study starts in August 2022 and ends in February 2023.

If you are in Group B, you will register on the Xiaoetong online learning platform after signing the informed consent, and then participate in a 7-month evidence-based leadership training program. The program will consist of 7 online modules, the training tutors will distribute reading materials to you through the Online Learning Platform, and you can study and complete the learning tasks on your own within the time period specified by researchers.

Compensation/Expenses: There will be no compensation for participation in this study, nor will there be any cost for you.

Risks: Participation in this study involves no risks to you.

Benefits: Participation in this study may improve your evidence-based leadership.

Alternatives: If you do not participate in this study, there are no alternatives other than work as usual, this study will not affect your work, and it will not affect your work.

Confidentiality: The information you provide will be kept strictly confidential (your name will not be recorded or shown in other research materials). We will number your data, and any information that identifies you will be obscured. Your name will not appear in the study results. Recorded interviews and related questionnaire data and materials will be stored on a USB stick and locked away from access by anyone other than the principal investigators.

Voluntary participation: You are free to choose to participate or not. If you participate, you can withdraw at any time for any reason. If you choose to withdraw from the project in the middle of the process, we will respect your wishes and destroy or not perform any analysis of your data, but only keep it together with the data of other participants.

Questions: If you have any questions about this research project, you can ask now. If you have any questions in the future, please contact principal investigator, Xianhong Li. Contact information: 18374961210.

I have read the content provided above and Xianhong LI (principal investigator) has explained the project to me and answered any questions I have asked. I have been informed of the possible risks and inconveniences of participating in this project and the possible benefits. I have also been informed of the measures available to me in addition to those provided by the project.

I understand that I have the choice to not participate in this program and that there will be no penalty or impact on my rights (such as how I am perceived by my leadership or colleagues) if I refuse to participate. I may also withdraw from this program at any time.

I understand my rights as a study subject. I volunteer to participate in this study. I understand what this study is about, why it is being conducted, and what it will do. I will receive an informed consent form that requires signature.

| Signature o | of the study | subject | |
|-------------|--------------|-----------|--------------------------|
| (Please sig | n if you ag | ree to pa | rticipate in this study) |
| Year | _ Month _ | _ Day | |

Signature of principal investigator or person administering informed consent:

Contact information: 18374961210

If you do not agree to participate in this study, please click "Disagree and Exit", if you agree to participate in this study, please click "Agree and Continue" to complete the baseline survey and submit it.

June 25, 2022

### 知情同意书

项目名称:循证领导力培训,提高护理领导者的领导力

项目负责人: 李现红, 博士, 中南大学湘雅护理学院教授; VÄLIMÄKI Maritta, 博 士,图尔库大学教授。

您将被邀请参加 循证领导力培训,提高护理领导者的领导力 研究项目。此项目的 目的是 为护理领导者领导力的干预提供切实可行的方案,以促进护理领导者领导 力的提升。

此项目将从 2022 年 08 月 2023 年 02 月实施, 共 7月。

## 如果您同意参加此项目:

- 1. 项目负责人将在您方便的时候对您进行访谈。
- 2. 您将有可能被问到有关 参与本项目次数及感受等 方面的问题。访谈将会被录 音, 访谈大概持续30分钟(在项目结束后的一周)。
- 3. 您将被要求填写一份问卷(共3次,项目开始前后各一次,项目结束7个月后一 次)。
- 4. 您有权在任何时刻以任何理由终止访谈。
- 5. 访谈结束后,作为感谢,您将收到一个有纪念意义的书签。

如果您在A组, 您将 在同意参与本研究后, 通过小鹅通在线学习平台进行注册, 然后参与为期7个月的循证领导力培训。本次培训为7次录课形式的线上课程,每月 一次,每次课程均围绕一个主题,持续30分钟左右,线上课程结束后将有对应课程 的课后训练和/或课后阅读材料(阅读材料包括PPT、文献资料、视频等),每个参 与者需在下次课程开始前完成本次课程的课后训练并上传至小鹅通,可在规定时间 内自主选择学习时间,如:第一次课程的课后训练为根据所学课程确定一个参与者 在自身工作中面临的领导力问题,并对其进行清晰的描述,然后将详细的问题在下 次课程开始前上传至学习通。研究从2022年8月开始,2023年2月结束。

如果您是在B组,您将 在同意参与本研究后,通过小鹅通在线学习平台进行注 册,然后参与为期7个月的循证领导力培训。本次培训为7次线上形式的培训,培训 导师将在小鹅通在线学习平台为您发放相关的阅读材料,您可以在规定时间自行学 习,并完成相应的学习任务。

## 补偿/花费

参加此项目将不会有任何补偿,也不会对您产生任何费用。

风险:参与此项目不会给您带来任何风险。

收益:参与此项目将可能促进您本人循证领导力的提升。

替代措施:如果不参与本研究,不存在替代方案,不会影响您的工作。

保密措施: 您所提供的信息我们将会严格保密(您的姓名将不会被录音或者出现在 其他研究材料上)。我们将对您的资料进行编号,任何可识别您身份的信息都会被 屏蔽。呈现研究结果时将不会出现您的名字。访谈录音和相关问卷数据与资料将被存放于U盘中并锁起来,除了项目负责人外,其他人均无法接触。

自愿参加:您可以自由选择参加或者不参加,如果您参加了,也可以在任何时刻以任何理由退出而不会影响到您的工作;如果您选择中途退出本项目,我们将尊重您的意愿,销毁或不对您的数据进行任何分析,而只是与其他参与者的数据一起保存。

疑问:关于此研究项目,如果您有任何疑问,现在可以提出。如果将来您还有什么问题,请联系项目负责人李现红,电话18374961210。

我已阅读上述所提供内容,李现红(项目负责人)已给我解释了此项目并回答了我 所提出的问题。我已被告知参与此项目可能存在的风险和不便之处及可能带来的好 处。我也被告知除项目所提供的措施外其他我可采用的措施。

我明白我可以不参加此项目,如果我拒绝参加将不会有任何惩罚或影响我应有的权利(如领导或同事对我的看法)。我也可以随时退出此项目。

我明白作为一个研究对象我该享有的权利。我自愿参加此研究。我明白此研究是干什么的,为什么要进行此研究以及将要怎么做。我将会收到一份需要签名的知情同意书。

| 研究对象签名 | (如您同意参 | 与本研究, | 请签名) |
|-----------|-----------------|-------|------|
| 年 | 月 日 | 1 | |
| 项目负责人或抗 | <b>执行知情同意</b> 者 | ¥签名: | |
| 联系方式: 183 | 74961210 | | |

如您不同意参与本研究,请点击"不同意并退出";如您同意参与本研究,请点击"同意并继续",完成学员基线调查并提交。

2022年6月25日